CLINICAL TRIAL: NCT03797339
Title: Multi-omics Study of the Individual Differences of Drug Efficacy and Toxicity in Patients With Coronary Heart Disease
Brief Title: Multi-omics Study of Clinical Endpoints in CHD
Acronym: OmiDETCHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: RenJi Hospital (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, ShiLong Zhong, Professor, Guangdong Provincial People's Hospital
Other Study IDs: 2017YFC0909301
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Coronary Heart Disease
Keywords: epigenome; metabolome; microbiome; genome; multi-omics targets; individual drug use
MeSH Terms: conditions — Coronary Disease | interventions — Validation Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces,urine,and blood are from patients with coronary heart disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discovery cohort: 1000 cases of coronary heart disease follow-up cohort was used for multi-omics target discovery.During the follow-up period, the information about the occurrence and risk factors of adverse cardiovascular events will be collected.
  Interventions: Other: risk factors of adverse cardiovascular events; Other: multi-omics target discovery
- Validation corhort: 3000 coronary heart disease follow-up cohorts was used for validating the results from the discovery corhort. During the follow-up period, the occurrence and risk factors of adverse cardiovascular events.Predictive mathematical models based on multi-omics combination will be constructed finally.
  Interventions: Other: risk factors of adverse cardiovascular events; Other: validation; Other: Predictive mathematical models

INTERVENTIONS:
Other: risk factors of adverse cardiovascular events — During the follow-up period,general information(age, sex, BMI, blood pressure, the history of drink and smoke, medical history, etc).Blood biochemistry parameters（Lipid, hsCRP levels, etc）and other laboratory examination parameters will be collected
Other: multi-omics target discovery — Genome-wide genotype , DNA methylation and metabolomes were determined using illumina high-density genotyping chips, high-throughput sequencing, and high-resolution mass spectrometry respectly. Blood exposure of statins and metoprolol and its metabolites was determined by UPLC-MS/MS.
  Groups: Discovery cohort
Other: validation — The genome-wide genotype of patients with coronary heart disease was detected using the illumina chip. The methylation level of the functional region was detected by the target region enrichment methylation sequencing method. Intestinal flora differences were detected using 16SrDNA high-throughput sequencing.
  Groups: Validation corhort
Other: Predictive mathematical models — Machine learning algorithms such as multiple linear regression or Bayesian classification are used to optimize clinical factors and multi-group targets to establish predictive mathematical models.
  Groups: Validation corhort

SUMMARY:
This study aimed to explore underlying mechanisms of individual differences in drugs for coronary heart disease treatment and its association with adverse consequences. It will enroll approximately 4000 coronal heart disease patients aged between 18 and 80 years in mainland China and follow-up for at least 1 years. Questionnaires, anthropometric measures, laboratory tests, and biomaterials will be collected . The principal clinical outcomes of the study consist of ischemia attack , cardiac death, renal injury,and myotoxic activity.

DETAILED DESCRIPTION:
The study is a multicenter prospective cohort study, aimed to explore underlying mechanisms of individual differences in drugs for coronary heart disease treatment and its association with adverse consequences.The genomic genotype, DNA methylation and metabolome of 1000 patients with coronary heart disease were determined using illumina high-density genotyping chip, high-throughput sequencing and high-resolution mass spectrometry. Blood exposures of statins and metoprolol and its metabolites was determined by UPLC-MS/MS.

The biological network using cross-omics analysis was reconstructed to identify potential causative key genes, bacteria, and endogenous metabolite targets that cause differences in individual responses. A machine identification algorithm selecting clinical factors and multi-omics targets was used to establish a predictive mathematical model.

A multi-center clinical cohort of 3000 coronal heart disease patients was used to verify the effects of various levels of omic targets on drug blood exposures, efficacy and toxic side effects. A comprehensive model based on multi-target combination of individualized drugs was constructed, and the predictive effect was clinically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-80 years
* Chinese Han patients with coronary artery disease
* inpatients undergoing coronary angiography or percutaneous coronary intervention

Exclusion Criteria:

* renal insufficiency (defined as serum creatinine concentration > 2 times the upper limit of normal [230 μmol/L], renal transplantation or dialysis)
* hepatic insufficiency (defined as serum transaminase concentration > 2 times the upper limit of normal [80 U/L], or a diagnosis of cirrhosis)
* pre-existing bleeding disorders
* being pregnant or lactating
* advanced cancer or haemodialysis
* history of thyroid problems, and use of antithyroid drugs or thyroid hormone medication
* incomplete information about cardiovascular events during follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Han patients with coronary artery disease who have ingested metoprolol and statins were prospectively recruited from Guangdong General Hospital, Shanghai Jiao Tong University, Central South University, Sun Yat-sen University and Sichuan University.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | from date of baseline examination until the date of first documented death,up to 48 months
  All-cause death

SECONDARY OUTCOMES:
MACE | from date of baseline examination until the date of first documented cardiovascular events,up to 48 months
  MACE was defined as the occurrence of cardiac death, nonfatal myocardial infarctions, coronary revascularisation and cerebral infraction.
Bleeding | from date of baseline examination until the date of first documented bleeding,up to 48 months
  Bleeding was the six-month incidence of combined alarming, internal, and nuisance bleeding events defined according to Serebruany et al15. Alarming bleeding included bleeding requiring a transfusion, intracranial bleeding, and life-threatening bleeding. Internal bleeding included haematoma, epistaxis, blood loss from the mouth, vagina, melaena, eye bleed, haematuria, and haematemesis. Nuisance bleeding included easy bruising, bleeding from small cuts, petechiae, and ecchymosis.
Statin-induced myopathy (SIM) | from date of baseline examination until the date of first documented SIM,up to 48 months
  The definition of SIM from statin treatment was based on the patients' subjective sense of muscular pain as well as CK elevations. These muscular side effects included myalgia (muscle pain/ache without serum CK elevations), other muscle-related symptoms such as weakness, cramps, spasms, soreness and twitching, CK elevations without physical symptoms, myositis or other muscle symptoms with CK elevations, and rhabdomyolysis.
CI-AKI | more than 6 h within 48 h after Coronary Angiography
  CI-AKI was diagnosed if a patient had an absolute increase in serum creatinine (sCr) concentration ≥ 0.3 mg/dl (26.4 μmol/L) from baseline or a relative increase ≥ 50 % in sCr concentration for more than 6 h within 48 h after surgery

OTHER OUTCOMES:
SYNTAX score | more than 6 h within 48 h after Coronary Angiography
  It is mainly used for the treatment of left main coronary artery lesions and/or three-vessel lesions.Patients with a score of ≥33 are recommended for CABG. Patients with a score between 23 and 32 can choose either PCI or CABG. Patients with a score of ≤22 are recommended for PCI and CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Shilong Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (5):
- China (5):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - XiangYa Hospital Central South University, Changsha, Hunan
  - Renji Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Derived] Chen Y, Jiang H, Zhan Z, Lu J, Gu T, Yu P, Liang W, Zhang X, Liu S, Bi H, Zhong S, Tang L. Restoration of lipid homeostasis between TG and PE by the LXRalpha-ATGL/EPT1 axis ameliorates hepatosteatosis. Cell Death Dis. 2023 Feb 6;14(2):85. doi: 10.1038/s41419-023-05613-6. PMID 36746922